CLINICAL TRIAL: NCT03670238
Title: Orogastric Intubation With Dental Fixation Versus Nasogastric Intubation: a Cross-over Randomized Trial
Brief Title: Orogastric Versus Nasogastric Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade de Passo Fundo (Other)
Responsible Party: Principal Investigator, Fernando Fornari, Clinical Professor, Universidade de Passo Fundo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Universidade de Passo Fundo
Record Dates: First submitted 2018-08-26; First posted 2018-09-13 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Feeding Patterns
Keywords: Nasogastric intubation; Orogastric intubation; Feeding tubes
MeSH Terms: conditions — Feeding Behavior | interventions — Intubation, Gastrointestinal

STUDY DESIGN:
Intervention Model Description: A cross-over randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orogastric intubation (Experimental): Orogastric intubation using a polyurethane enteral tube followed by fixation of the tube tip to a superior molar.
  Interventions: Device: Orogastric intubation
- Nasogastric intubation (Active Comparator): Nasogastric intubation using a polyurethane enteral tube followed by fixation of the tube to the patient face.
  Interventions: Device: Nasogastric intubation

INTERVENTIONS:
Device: Orogastric intubation — Patient was placed in Fowler position (45º) and intraoral infiltrative anesthesia was carried out with Lidocaine 2% (without vasoconstrictor) at gingival papilla in the vestibular-palatine direction. A polyurethane enteral tube (Medicone®, Cachoeirinha - Brazil) was inserted through the mouth and passed into de stomach, followed by fixation of the tube tip to a superior molar or premolar, in its palatine surface. For dental amarry it waas used a suture wire in stainless steel size 1.0
  Arms: Orogastric intubation
Device: Nasogastric intubation — After nostril anesthesia with xylocaine gel, a polyurethane enteral tube was inserted through the nose and its tip was positioned in the gastric lumen, according to the nose-ear-xiphoid method. The tube was attached to the face using antiallergic adhesive tape.
  Arms: Nasogastric intubation

SUMMARY:
Feeding by tube is commonly used for inpatients and ambulatory patients. For this purpose nasogastric (NG) intubation is the traditional approach. The aim of this study was to develop the orogastric (OG) intubation with dental fixation and compare OG versus NG intubation in healthy volunteers.

DETAILED DESCRIPTION:
In this randomized, open label, clinical trial with crossing over design, 13 healthy individuals were invited to participate. The study was performed at Hospital São Vicente de Paulo between July and December 2017. Those who accepted were studied after signing an informed consent form. Sample estimation (software WinPEPI) indicated that 13 participants would be enough to show a difference between OGI and NGI of 1 hour in terms of tolerance (SD 30 min), with alpha 5% and power of 80%. Inclusion criteria were age between 18 and 70 years, absence of any acute or chronic disease and intact upper posterior molars or premolars. The study was conducted according to rules of the Helsinki declaration and was approved by the local Ethical Committee (number 1.942.505).

The participants were randomly allocated to OG and NG intubations with a 15 days interval. Randomization was carried out with computed generated aleatory numbers. A trained dentist (RS) performed OG intubation with dental fixation. After explanation about the procedure, the patient was placed in Fowler position (45º) and intraoral infiltrative anesthesia was carried out with Lidocaine 2% (without vasoconstrictor) at gingival papilla in the vestibular-palatine direction. A polyurethane enteral tube (Medicone®, Cachoeirinha - Brazil) was inserted through the mouth and passed into de stomach, followed by fixation of the tube tip to a superior molar or premolar, in its palatine surface. For dental amarry we used a suture wire in stainless steel size 1.0 (Johnson & Johnson - Ethicon, São Paulo, Brazil).

NG intubation followed the traditional steps described elsewhere and was executed by the first author (RS). Briefly, after nostril anesthesia with xylocaine gel, a polyurethane enteral tube was inserted through the nose and its tip was positioned in the gastric lumen, according to the nose-ear-xiphoid method. The tube was attached to the face using antiallergic adhesive tape.

During both OG and NG intubations the participants were monitored regarding the occurrence of nausea, vomit, cyanosis, dyspnea, cough and discomfort. A bottle containing 900 ml of enteral diet (1.5kcal/ml, Nutrison Energy - Danone®, São Paulo - Brazil) was provided for each participant, with instructions of use. They were explained how to manually remove the tube if necessary, and asked to return to the hospital in the following day.

The main efficacy outcome was tolerance in hours. After intubation patients were asked to return in 24 hours for tube removal, but were allowed to withdraw the tube at any time in case of substantial discomfort. Secondary outcomes were discomfort, handling, speech, mastication, deglutition and esthetic. These efficacy outcomes were assessed using a self-reporting questionnaire in which participants were asked to reply after tube removal. Each outcome was rated by means of a 10-item Likert scale (0 = best / 10 = worst). Safety outcomes were registered either by the researcher during the intubation procedure (placement and removal) or by the participants replying an open question: "please describe any complaint related with the intubation".

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years;
* Healthy volunteers;
* Individuals to participate in the study who referred to becoming superior of the subsequent intact students (Molars or premolars, either side);
* Individuals of both sexes.

Exclusion Criteria:

* Gastroesophageal complaints;
* Limitation of mouth opening;
* Pathologies of airways;
* Individuals invited to the study who reported bilateral upper posterior tooth loss;
* Inability to respond to the questionnaire

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08-10 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-12-10 (Actual)

PRIMARY OUTCOMES:
Tolerance | two days
  Period in hours (maximum 24 hours) that the patients tolerated the intubation, ranging from zero to 24 hours.

SECONDARY OUTCOMES:
Discomfort | two days
  Patients will rate nose, oral and/or throat discomfort during nasogastric and orogastric intubation, according to a Likert scale, which ranges between 0 (no discomfort, better outcome), 1,2,3,4,5,6,7,8,9 and 10 (maximum discomfort, worse outcome), after each intubation. The intubations scores will be compared with paired t test.
Handling | two days
  Patients will rate handling between 0 (worst) and 10 (best) after each intubation.
Speech | two days
  Patients will rate speech impairment during nasogastric and orogastric intubation, according to a Likert scale, which ranges between 0 (no impairment, better outcome), 1,2,3,4,5,6,7,8,9 and 10 (maximum impairment, worse outcome), after each intubation. The intubations scores will be compared with paired t test.
Esthetic | two days
  Patients will rate esthetic impairment during nasogastric and orogastric intubation, according to a Likert scale, which ranges between 0 (no impairment, better outcome), 1,2,3,4,5,6,7,8,9 and 10 (maximum impairment, worse outcome), after each intubation. The intubations scores will be compared with paired t test.
Deglutition | two days
  Patients will rate deglutition impairment during nasogastric and orogastric intubation, according to a Likert scale, which ranges between 0 (no impairment, better outcome), 1,2,3,4,5,6,7,8,9 and 10 (maximum impairment, worse outcome), after each intubation. The intubations scores will be compared with paired t test.
Mastication | two days
  Patients will rate mastication impairment during nasogastric and orogastric intubation, according to a Likert scale, which ranges between 0 (no impairment, better outcome), 1,2,3,4,5,6,7,8,9 and 10 (maximum impairment, worse outcome), after each intubation. The intubations scores will be compared with paired t test.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Fornari, Professor, Study Director — Universidade de Passo Fundo
Locations (1):
- Renato dos Santos, Passo Fundo, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dos Santos R, Della Bona A, Fornari F. Orogastric intubation with dental fixation for enteral nutrition: a proof-of-concept study. Br J Oral Maxillofac Surg. 2021 Jul;59(6):672-677. doi: 10.1016/j.bjoms.2020.08.098. Epub 2020 Aug 25. PMID 33985848